CLINICAL TRIAL: NCT05486195
Title: A First-in-Human, Randomized, Placebo-controlled, Single Ascending Oral Dose Study of SDI-118 in Healthy Male Subjects Including Receptor Occupancy Measurements After Single Dose of SDI-118 and an Assessment of Food Effect
Brief Title: A Single Ascending Oral Dose Study of SDI-118 in Healthy Male Subjects Including an Assessment of Receptor Occupancy and Food Effect
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Syndesi Therapeutics (Industry); KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: SYND001; 2018-004022-28 (EudraCT Number)
Record Dates: First submitted 2022-08-02; First posted 2022-08-03 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Cognitive Disorders
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- SDI-118 Dose 1 (Experimental)
  Interventions: Drug: SDI-118
- SDI-118 Dose 2 (Experimental)
  Interventions: Drug: SDI-118
- SDI-118 Dose 3 (Experimental)
  Interventions: Drug: SDI-118
- SDI-118 Dose 4 (Experimental)
  Interventions: Drug: SDI-118
- SDI-118 Dose 5 (Experimental)
  Interventions: Drug: SDI-118
- SDI-118 Dose 6 (Experimental)
  Interventions: Drug: SDI-118
- SDI-118 Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SDI-118 — SDI-118 Powder in Capsule
  Arms: SDI-118 Dose 1; SDI-118 Dose 2; SDI-118 Dose 3; SDI-118 Dose 4; SDI-118 Dose 5; SDI-118 Dose 6
Drug: Placebo — Matching Placebo
  Arms: SDI-118 Placebo

SUMMARY:
This is a First-in-Human, Randomized, Placebo-controlled, Single Ascending Oral Dose Study of SDI-118 in Healthy Male Subjects including Receptor Occupancy Measurements after Single Dose of SDI-118 and an Assessment of Food Effect.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects, 18 to 50 years of age, inclusive.
* Non-smokers or abstinence from tobacco for at least 3 months prior to screening.
* Body mass index (BMI) between 18 and 30 kg/m2, inclusive, with a minimum weight of 50 kg and maximum of 100 kg.
* Venous access sufficient to allow blood sampling as per the protocol.
* Agree to abstain from alcohol intake 24h before each administration of study drug, during the in-patient period of the study and 24 hours prior to all other out-patient clinic visits.
* Have given written informed consent approved by the relevant Ethics Committee (EC) governing the site.
* In the Investigator's opinion, subject is able to understand the nature of the study and any risks involved in participation, and willing to cooperate and comply with the clinical study protocol restrictions and requirements.
* Subjects and their partners of childbearing potential must be willing to use 2 methods of contraception, one of which must be a barrier method, for the duration of the study and up to 90 days after the last dose.

Specifically, Part B/PET related inclusion criteria:

* Adequate arterial circulation in both hands (Allen's test).
* MRI scan without clinically significant abnormalities.

Specifically, Part C/FE related inclusion criteria:

* Subjects are not vegetarian and willing to eat a standardized high fat breakfast including butter and bacon.

Exclusion Criteria:

* History or symptoms of any significant disease including (but not limited to), neurological, psychiatric, endocrine, cardiovascular, respiratory, gastrointestinal (GI), hepatic, or renal disorder.
* Positive Hepatitis B surface antigen (HBs Ag), Hepatitis C antibody (HCV Ab), or human immunodeficiency virus antibody (HIV Ab) at screening.
* Use of any medications (prescription or over-the-counter (OTC)), vitamin, mineral, herbal, and dietary supplements (including grapefruit products) within 7 days of study drug administration, or less than 5 half-lives (whichever is longer).
* Have an estimated Glomerular Filtration Rate (eGFR) <80 mL/min/1.73m2.

Any of the following findings in the resting ECG:

* QTcF> 450 or < 300 msec at screening or baseline visit,
* Notable resting bradycardia (HR < 40 bpm) or tachycardia (HR > 100 bpm) at screening or baseline visit,
* Personal or family history of congenital long QT syndrome or sudden death,
* Screening or baseline ECG with QRS and/or T wave judged to be unfavourable for a consistently accurate QT measurement (e.g. neuromuscular artefact that cannot be readily eliminated, arrhythmias, indistinct QRS onset, low amplitude T wave, merged T- and U-waves, prominent U waves),
* Evidence of atrial fibrillation, atrial flutter, Left Bundle Branch Block (LBBB), Wolf-Parkinson-White Syndrome, or cardiac pacemaker at screening or baseline visit (note: a first degree heart block with PR not exceeding 250 msec can be allowed).

Specifically, Part B/PET related exclusion criteria:

* Previous inclusion in a research study and/or medical protocol involving nuclear medicine, PET or radiological investigations with significant radiation burden (a significant radiation burden being defined as International Commission on Radiological Protection (ICRP) category IIb or above: no more than 1 mSv in addition to the natural background radiation in the previous 12 months including the dose from the study).
* Subject who fulfils any of the MRI contraindications on the standard radiography screening questionnaire (including the presence of ferromagnetic metal in the body or heart pacemaker).
* History of or suffers from claustrophobia or feels that they will be unable to lie still on their back in the PET camera for a period of 2 hours.
* Any known allergy to local anaesthetics or heparin.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 32 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2019-07-29 (Actual); Study Completion 2020-03-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) | 21 Days
  Adverse events (AEs) will be coded using medical dictionary for regulatory activities (MedDRA). An AE is any untoward medical occurrence in a participant administered a study drug and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medical product whether or not considered related to the medical product. An AE is considered "serious" if, in the view of either the investigator or sponsor, the event: results in death, is life-threatening, results in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, results in congenital anomaly or birth defect, requires hospitalization or prolongation to hospitalization, or other medically important event.
Number of participants with laboratory value abnormalities and/or adverse events (AEs) | 21 Days
  Number of participants with potentially clinically significant laboratory values (hematology/chemistry/urinalysis)
Number of participants with vital sign abnormalities and/or adverse events (AEs) | 21 Days
  Number of participants with potentially clinically significant vital sign values
Number of participants with temperature abnormalities and/or adverse events (AEs) | 21 Days
  Number of participants with potentially clinically significant temperature values
Number of participants with routine 12 lead electrocardiogram (ECG) abnormalities and/or Adverse Events (AEs) | 21 Days
  Number of participants with potentially clinically significant ECG values.
Number of participants with routine physical examination abnormalities and/or Adverse Events (AEs) | 21 Days
  Number of participants with potentially clinically significant changes in physical examination.
Number of participants with routine neurological examination abnormalities and/or Adverse Events (AEs) | 21 Days
  Number of participants with potentially clinically significant changes in neurological examination.
Number of participants with abnormalities on Profile of Mood States (Brief) and/or Adverse Events (AEs) | 21 Days
  Number of participants with potentially clinically significant changes in Profile of Mood States (Brief) values.
Number of participants with abnormalities on Bond-Lader-VAS and/or Adverse Events (AEs) | 21 Days
  Number of participants with potentially clinically significant changes in Bond-Lader VAS values.

CONTACTS AND LOCATIONS:
Overall Officials: Jan deHoon, MD, Principal Investigator — UZ Leuven
Locations (1):
- Centre for Clinical Pharmacology, UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Botermans W, Koole M, Van Laere K, Savidge JR, Kemp JA, Sunaert S, Duffy MM, Ramael S, Cesura AM, D'Ostilio K, Gossen D, Madsen TM, Lodeweyckx T, de Hoon J. SDI-118, a novel procognitive SV2A modulator: First-in-human randomized controlled trial including PET/fMRI assessment of target engagement. Front Pharmacol. 2023 Jan 17;13:1066447. doi: 10.3389/fphar.2022.1066447. eCollection 2022. PMID 36733374